CLINICAL TRIAL: NCT04548349
Title: Profiling the Skin Microbiome in Response to Altreno in Acne Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Ortho Dermatologics (Industry)
Responsible Party: Principal Investigator, Jean S. McGee, MD, PhD, Assistant Professor of Dermatology, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P000595
Record Dates: First submitted 2020-07-20; First posted 2020-09-14 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Acne; Healthy
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin; Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Altreno Group (Experimental)
  Interventions: Drug: Altreno
- BPO Group (Experimental)
  Interventions: Drug: Benzoyl peroxide
- Control Group (No Intervention): During the entire study period, the subjects in the control group will not be allowed to use any antibacterial wash, other than approved OTC cleansers.

INTERVENTIONS:
Drug: Altreno — Acne patients will be assigned to Altreno once daily.
  Arms: Altreno Group
Drug: Benzoyl peroxide — Acne patients will be assigned to BPO leave-on gel once daily.
  Arms: BPO Group

SUMMARY:
The study objective is to characterize the shift in the diversity and abundance of the skin microbial community at baseline and in response to Altreno monotherapy as compared to benzoyl peroxide (BPO) 2.5% leave-on gel monotherapy in acne patients.

DETAILED DESCRIPTION:
With the advent of 16S rRNA sequencing, scientific community is beginning to understand the critical importance of the microbiome in human health. In dermatology, researchers have begun to lead the effort to not only better understand how the microbiome contributes to the pathogenesis of skin disease, but also harness its power to develop novel therapies. Acne is a common inflammatory skin disorder. P. acnes on the skin has been traditionally thought of as the culprit bacteria in the pathogenesis of acne.

Recent studies demonstrate that the skin microbial composition dynamically changes in response to systemic acne therapy. Using 16 rRNA gene sequencing, a prior study has confirmed that systemic antibiotic treatment decreased the abundance of P. acnes, which returned to baseline after discontinuation of the therapy. In contrast, the systemic therapy increased the abundance of Pseudomonas species, which returned to baseline after therapy cessation. Based on the opposing response to the therapy, it can be speculated that these two species compete for the same microenvironment within the skin microbiome. Interestingly, the same systemic therapy decreased the abundance of lactobacillus genus, the "good bacteria" that is protective against skin infection, and that decrease was sustained even after cessation of the therapy. Similarly, another study has demonstrated that systemic isotretinoin therapy disturbed the skin microbiome in acne patients with increased bacterial diversity on the cheeks. It is unclear the potential therapeutic role of the increased bacterial diversity in the management of acne patients.

The study aims to characterize the shift in the diversity and abundance of the skin microbial community in response to Altreno in acne patients. Understanding the role of the skin microbiome in response to therapy can help clinicians to develop tailored, targeted treatment options, including reconstitution of "good bacteria." Furthermore, it can lead to development of novel topical pre and probiotics.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of acne that warrants initiating topical medications.
* Denies use of any prescribed systemic acne treatments in the past 30 days.
* Denies use of any prescribed topical medications in the past 30 days.
* Denies use of any OTC topical acne medications in the past 14 days.
* Denies use of any emollients in the past 24 hours (if feasible).
* Denies bathing or facial washing in the past 12 hours (if feasible).
* Willingness to adhere to the recommended topical regimen during the duration of the study.

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to get pregnant during the study.
* Use of any investigational drug(s) in the past 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deacones Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Chien AL, Tsai J, Leung S, Mongodin EF, Nelson AM, Kang S, Garza LA. Association of Systemic Antibiotic Treatment of Acne With Skin Microbiota Characteristics. JAMA Dermatol. 2019 Apr 1;155(4):425-434. doi: 10.1001/jamadermatol.2018.5221. PMID 30758497
- [Background] Kelhala HL, Aho VTE, Fyhrquist N, Pereira PAB, Kubin ME, Paulin L, Palatsi R, Auvinen P, Tasanen K, Lauerma A. Isotretinoin and lymecycline treatments modify the skin microbiota in acne. Exp Dermatol. 2018 Jan;27(1):30-36. doi: 10.1111/exd.13397. Epub 2017 Sep 14. PMID 28636791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The BPO arm was not included in this reporting. We only recruited 1 subject in this arm and did not reach the sufficient number needed to make meaningful comparisons. It was decided that we would proceed with comparing no acne vs. acne treated with Altreno. We did not pursue any downstream processing of the samples collected from that 1 patient, so no results are available for this arm. ***The BPO Arm, 1 subject enrolled, but no analysis formed.***
Groups:
- Altreno Group: Altreno (0.05% lotion): Acne patients will be assigned to Altreno once daily.
- BPO Group: BPO 2.5% leave-on gel: Acne patients will be assigned to BPO once daily.
Period: Overall Study
Arm/Group | Altreno Group | Control Group | BPO Group
Started | 12 | 12 | 1
Completed | 8 | 8 | 1
Not Completed | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Population: As described in the Pre-Assignment Details section, BPO arm was excluded from the study. We did not pursue processing the samples from 1 recruited subject in this arm. Therefore, we do not have any results to report.
Groups:
- BPO Group: BPO: Acne patients will be assigned to BPO once daily.
- Total: Total of all reporting groups
Arm/Group | Altreno Group | Control Group | BPO Group | Total
Number analyzed (Participants) | 12 | 12 | 1 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (6.4) | 31.8 (4.9) | 26 (0) | 30.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 1 | 18
  Male | 1 | 6 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 11 | 11 | 1 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 9 | 12 | 1 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Relative Abundance [Median (Inter-Quartile Range); unit: Relative Abundance] — We are not reporting the baseline relative abundance for the overall population. The relative abundance is calculated for control group and for acne group separately. Because the outcome measure that we are looking for is the change from the baseline relative abundance after intervention within each group, not as the overall population. Population: We are not reporting the baseline relative abundance for the overall population. The relative abundance is calculated for control group and for acne group separately. Because the outcome measure that we are looking for is the change from the baseline relative abundance after intervention within each group, not as the overall population.
  Relative Abundance
    Altreno Group: number analyzed (Participants) | 12 | 0 | 0 | 12
    Altreno Group | 3.29 [2.38 to 5.32] |  |  | 3.29 [2.38 to 5.32]
    Control Group: number analyzed (Participants) | 0 | 12 | 0 | 12
    Control Group |  | -2.49 [-3.24 to -2.19] |  | -2.49 [-3.24 to -2.19]

OUTCOME MEASURES:

1. Primary Outcome: CLR-transformed Abundance of Any Significant Taxa
Description: The primary outcome measures the relative abundance of Kingella after treatment with Altreno in acne patients vs without treatment in healthy subjects. The relative abundance was represented as centered log ratio (CLR) transformation. These values are all relative terms centered around 0, more negative means less abundant in comparison. More positive means more abundant in comparison.
Time Frame: Baseline, 90 days after treatment, and followed by 30 days of no treatment
Population: The participants analyzed differ because of lost to follow-up and/or not sufficient DNA yield for downstream microbiome sequencing.
Measure: Median (Inter-Quartile Range); unit: Relative Abundance
Arm/Group | Altreno Group | Control Group
Number analyzed (Participants) | 11 | 10
Relative Abundance
  Baseline | 3.29 [2.38 to 5.32] | -2.49 [-3.24 to -2.19]
  +90 days from baseline: number analyzed (Participants) | 8 | 6
  +90 days from baseline | -1.59 [-2.98 to 1.88] | -2.75 [-2.92 to -2.21]
  +120 days from baseline: number analyzed (Participants) | 11 | 0
  +120 days from baseline | -1.98 [-3.51 to 3.37] |

ADVERSE EVENTS:
Time Frame: The adverse events were asked at each study visit. For both groups, adverse events were collected over ~120 days.
Groups:
- Altreno Group: Altreno 0.05% lotion: Acne patients will be assigned to Altreno once daily.
- BPO Group: BPO 2.5% leave-on gel: Acne patients will be assigned to once or twice daily as tolerated.
Arm/Group | Altreno Group | Control Group | BPO Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/1
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/1

LIMITATIONS AND CAVEATS:
* BPO arm only have 1 participant, so we decided to drop this arm.
* Small sample size, high drop out rate, and high failure rate of DNA extraction were the limitations of this study among others.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT04548349/Prot_SAP_001.pdf